CLINICAL TRIAL: NCT06561009
Title: Safety and Efficacy of BAFFR CART for Relapsed/ Refractory Neuromyelitis Optica Spectrum Disorder
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Qiang Liu, Department of Neurology, Tianjin Medical University General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB2024-YX-220-01
Record Dates: First submitted 2024-07-23; First posted 2024-08-19 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Neuromyelitis Optica Spectrum Disorder
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant Group (Experimental): BAFFR CART cells
  Interventions: Drug: Anti-BAFFR CART

INTERVENTIONS:
Drug: Anti-BAFFR CART — Anti-BAFFR CART

SUMMARY:
This is an open-label, single-arm, dose-escalation study in up to 20 participants with relapsed/refractory Neuromyelitis Optica Spectrum Disorders (NMOSD). The aim is to evaluate the safety and efficacy of the treatment with BAFFR CART.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18-60 years;
2. Patients must be diagnosed as AQP4-IgG-positive NMOSD;
3. At least one immunosuppressant has been used for over a year with poorly controlled symptoms;
4. Clinical evidence of at least two relapses in the last 12 months or three relapses in the last 24 months and one relapse in the preceding 12 months before screening.
5. Subjects and their partners must be willing to use effective and reliable methods of contraception, devices or medicines, within one year before BAFFR CART cells infusion.
6. Subjects must provide written informed consent before the study begins and comply with the requirements of the study protocol.

Exclusion Criteria:

1. Subjects have received B cell deletion treatment within 6 months before screening;
2. Chronic and active hepatitis B (HBV), hepatitis C (HCV), Human Immunodeficiency Virus (HIV) infection, CMV or syphilis infections concurrently.
3. Subjects with Papovaviruses infection.
4. Subjects have received live attenuated vaccine vaccination within 8 weeks before screening; or plan to receive live vaccine vaccination within 8 weeks after treatment;
5. History of psychoactive drug abuse and failed to withdraw, or have a history of psychiatric disorders.
6. Pregnant or lactating women.
7. Subjects with severe heart, liver, kidney or bone marrow function disorder.
8. Allergic constitution or a history of severe allergies.
9. Subjects with conditions adjudicated by the investigator as unsuitable for lymphodepletion or cell infusion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) | Up to 28 days
  Incidence of dose-limiting toxicity (DLT) will be evaluated within the first 28 days following BAFFR CART cells infusion.
Incidence and severity of adverse events | Up to 28 days
  Adverse events will be evaluated following the chemotherapy preparative regimen and infusion of BAFFR CART cells within the first 28 days.

SECONDARY OUTCOMES:
Proportion of BAFFR CART cells in peripheral blood | Up to 1 years
  The proportion of BAFFR CART cells in peripheral blood will be detected after infusion.
Annualized relapse rate (ARR) | Up to 1 years
  ARR is defined as the number of attacks divided by the total participant-years after infusion.
Changes of B cell levels in bone marrow and peripheral blood | Up to 1 years
  The changes of B cell levels in bone marrow and peripheral blood after BAFFR CART infusion.
Changes of AQP4 antibody titers | Up to 1 years
  Changes of AQP4 antibody titers from baseline over 1 year after BAFFR CART infusion.
Changes of cytokine in peripheral blood | Up to 1 years
  Changes of cytokine(including IL-6, IFN-γ, TNF-α, and serum BAFF) in peripheral blood from baseline over 1 year after BAFFR CART infusion.
Changes of Expanded Disability Status Scale (EDSS) score | Up to 1 years
  Participant will be considered to have a worsening in overall EDSS score of at least 2 if baseline EDSS score was 0, or at least 1 point if baseline EDSS score is 1 to 5, or at least 0.5 point if baseline EDSS score is 5.5 or more.
Changes of visual acuity | Up to 1 years
  Corrected visual acuity is determine by Snellen E chart held at a distance of 5 meters.
Accumulated total active MRI lesions | Up to 1 years
  The changes of T2 lesions and/or enhancing T1 Lesions as detected by brain Magnetic Resonance Imaging (MRI).